CLINICAL TRIAL: NCT06638840
Title: Pediatric Performance and Satisfaction of Oticon Medical Ponto on Softband.
Status: Completed | Type: Observational
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: BC117
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study is a non-interventional, observational, study on users of Ponto sound processors who use their sound processors on a softband solution. The purpose of this study is to assess subjective benefit by evaluating performance and overall satisfaction of the Ponto on a Ponto Softband in pediatric users.

ELIGIBILITY:
Inclusion Criteria:

* currently using Oticon Medical Ponto sound processor on Oticon Medical Softband

Exclusion Criteria:

* not

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ponto sound processor users
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oticon Medical, Somerset, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants: Participants who participated in the survey (one armed study)
Period: Overall Study
Arm/Group | Participants
Started | 64
Completed | 47
Not Completed | 17

BASELINE CHARACTERISTICS:
Population: All 64 participants who participated in the survey
Arm/Group | Participants
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.0 (4.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 35
  Gender: Female | 28
  Gender: Do not wish to say | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: PEACH Overall Score
Description: Overall score from the Parents' Evaluation of Aural/Oral Performance of Children questionnaire (PEACH questionnaire). PEACH score is calculated as percentage of the maximum score (thus score is on a scale of 0-100%). Higher score indicate better performance.
Time Frame: Single timepoint for completion of survey
Population: Full analysis set of all participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Participants
Number analyzed (Participants) | 64
Score on a scale | 76.1 (14.4)

2. Primary Outcome: Quiet PEACH
Description: Quiet score from the Parents' Evaluation of Aural/Oral Performance of Children questionnaire (PEACH questionnaire). PEACH score is calculated as percentage of the maximum score (thus score is on a scale of 0-100%). Higher score indicate better performance.
Time Frame: Single timepoint for completion of survey
Population: Full analysis set of all participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Participants
Number analyzed (Participants) | 64
Score on a scale | 81.0 (12.8)

3. Primary Outcome: Noise PEACH
Description: as for outcome 1
Time Frame: Single timepoint for completion of survey
Population: Full analysis set of all participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Participants
Number analyzed (Participants) | 64
Score on a scale | 70.3 (18.0)

4. Primary Outcome: Total GCBI Score
Description: Total score on the Glasgow Childrens Benefit Inventory (GCBI) questionnaire. Score is calculated on a scale of -100 to +100. The higher the score, the more benefit.
Time Frame: Single time point for completing survey
Population: Out of the 64 participants, only 47 completed the GCBI questionnaire.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Participants
Number analyzed (Participants) | 47
Score on a scale | 38.6 (27.4)

5. Primary Outcome: Psycho Social GCBI Score
Description: Psycho social score on the Glasgow Childrens Benefit Inventory (GCBI) questionnaire. Score is calculated on a scale of -100 to +100. The higher the score, the more benefit.
Time Frame: Single timepoint for completion of survey
Population: Out of the 64 participants, only 47 completed the GCBI questionnaire.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Participants
Number analyzed (Participants) | 47
Score on a scale | 27.9 (42.9)

6. Primary Outcome: Physical Health GCBI Score
Description: Physical health score on the Glasgow Childrens Benefit Inventory (GCBI) questionnaire. Score is calculated on a scale of -100 to +100. The higher the score, the more benefit.
Time Frame: Single timepoint for completion of survey
Population: Out of the 64 participants, only 47 completed the GCBI questionnaire.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Participants
Number analyzed (Participants) | 47
Score on a scale | 24.0 (13.3)

7. Primary Outcome: Behavior GCBI Score
Description: Behavior score on the Glasgow Childrens Benefit Inventory (GCBI) questionnaire. Score is calculated on a scale of -100 to +100. The higher the score, the more benefit.
Time Frame: Single timepoint for completion of survey
Population: Out of the 64 participants, only 47 completed the GCBI questionnaire.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Participants
Number analyzed (Participants) | 47
Score on a scale | 61.0 (34.5)

8. Primary Outcome: Vitality GCBI Score
Description: Vitality score on the Glasgow Childrens Benefit Inventory (GCBI) questionnaire. Score is calculated on a scale of -100 to +100. The higher the score, the more benefit.
Time Frame: Single timepoint for completion of survey
Population: Out of the 64 participants, only 47 completed the GCBI questionnaire.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Participants
Number analyzed (Participants) | 47
Score on a scale | 37.8 (30)

9. Primary Outcome: Use of Sound Processor
Description: Survey question: "Think about how much your child used their sound processor(s) over the past two weeks. On an average day, how many hours did they use the sound processor(s)?"
Time Frame: Single timepoint for completion of survey
Population: Full analysis set of participants
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 64
Participants
  Less than 1 hour | 1
  1 to 4 hours | 4
  4 to 8 hours | 15
  More than 8 hours | 43
  None | 1

10. Primary Outcome: Hearing Benefit
Description: Survey question: "Think about a situation where your child wanted to hear better, before receiving their sound processor. Over the past two weeks, how much has the sound processor(s) helped in that situation?"
Time Frame: Single timepoint for completion of survey
Population: Full analysis set of
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 64
Participants
  Helped not at all | 0
  Helped slightly | 3
  Helped moderately | 11
  Helped quite a lot | 14
  Helped very much | 35
  Not answered | 1

11. Primary Outcome: Overall Satisfaction - Ponto Experience
Description: Survey question: "How satisfied overall are you with your child's Ponto experience?"
Time Frame: Single timepoint for completion of survey
Population: Full analysis set of 64 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 64
Participants
  Very much | 37
  Quite a lot | 12
  Moderately | 13
  Slightly | 1
  Not at all | 1

12. Primary Outcome: Satisfaction With Softband
Description: Survey question: "How satisfied overall are you with your child's softband?"
Time Frame: Single timepoint for completion of survey
Population: Full analysis set of participants
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 64
Participants
  Very much | 14
  Quite a lot | 22
  Moderately | 18
  Slightly | 5
  Not at all | 5

ADVERSE EVENTS:
Time Frame: The study is a survey and did not include adverse event assessment
Description: The study is a survey and did not include adverse event assessment
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT06638840/Prot_SAP_000.pdf